CLINICAL TRIAL: NCT06812338
Title: Effect of Different Positions During Traction on Pain, Function, and Range of Motion in Adults with Non-specific Low Back Pain
Brief Title: Effects of Different Positions on Mechanical Traction Outcome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mshari Saleh Alghadier, Assistant Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT/024/020
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Non-specific Low Back Pain; Lumbar Traction

STUDY DESIGN:
Intervention Model Description: It will be a triple-armed Randomized control trial, 30 subject will be recruited and randomly allocated into the three groups (supine, prone, and side-lying) using sealed envelope method, same treatment will be delivered with difference in positioning only, Supine Participants will lie in supine position with legs supported on a stool adjusted for hip and knee flexion to be at 90°, Prone Participants will lie in prone position with a pillow underneath their abdomen and a harness attached to the chest, and pelvis. Side-lying Participants will lie on the contralateral side of pain, with his hip flexed at 80°, and a pillow between his knees.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Supine Participants (Active Comparator): Participants will lie in supine position with legs supported on a stool adjusted for hip and knee flexion to be at 90°
  Interventions: Device: mechanical traction
- Prone Participants (Active Comparator): will lie in prone position with a pillow underneath their abdomen and a harness attached to the chest, and pelvis
  Interventions: Device: mechanical traction
- Side-lying Participants (Active Comparator): will lie on the contralateral side of pain, with his hip flexed at 80°, and a pillow between their knees
  Interventions: Device: mechanical traction

INTERVENTIONS:
Device: mechanical traction — Participants will receive traction therapy as follows: force will start at 25% of Body weight, gradually increasing until the tolerance for pulling is reached with maximum of 50% of body weight. The session will be 15 minutes long (1min for acceleration, 13 min application, 1min deceleration); it will be intermittent with ratio of 30 s on and 10s off

SUMMARY:
Our primary purpose for this study is to investigate the effect of different positions during traction on pain, function, and range of motion in adults with non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-65 years of age
* Non specific LBP persisted for more than 12 weeks
* At least 4/10 on NPRS

Exclusion Criteria:

* Vertebral fractures
* Axial spondylarthritis
* Aauda equina syndrome
* Radicular pain
* Radiculopathy
* Spinal stenosis
* Spinal surgeries
* Malignancy
* Pregnancy
* Inflammatory or infectious cases of LBP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Arabic version | from baseline to the end of the 6th week
  assesses the impact of back pain on daily life across 10 sections. Each section covers different activities and aspects of daily living. The responses are scored from 0 (no impact) to 5 (maximum impact), with higher scores indicating greater disability

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) arabic version | from baseline to the end of the 6th week
  the questionnaire includes questions about various domains of activity, such as job-related activity, transportation, housework, and leisure-time physical activity
Numerical pain rating scale (NPRS) | from baseline to the end of the 6th week
  An 11-point scale that start at 0 (no pain) to 10 (worst imaginable pain)
Finger-to-floor test (FFT) | from baseline to the end of the 6th week
  Participants will be asked to bend forward as much as possible, the distance between the tip of the middle finger and the platform is measured in Cm using a measurement tape.

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided upon request through the principal investigator's email.

REFERENCES:
- [Background] Beattie PF, Nelson RM, Michener LA, Cammarata J, Donley J. Outcomes after a prone lumbar traction protocol for patients with activity-limiting low back pain: a prospective case series study. Arch Phys Med Rehabil. 2008 Feb;89(2):269-74. doi: 10.1016/j.apmr.2007.06.778. PMID 18226650
- [Background] Tanovic E, Celik D, Omerovic D, Zovko Omeragic V, Jaganjac A, Konjo H, Rovcanin E, Omerovic H. Intermittent traction therapy in the treatment of chronic low back pain. Med Glas (Zenica). 2021 Feb 1;18(1):158-163. doi: 10.17392/1252-21. PMID 33269579
- [Background] Yorkin M, Spaccarotella K, Martin-Biggers J, Quick V, Byrd-Bredbenner C. Accuracy and consistency of weights provided by home bathroom scales. BMC Public Health. 2013 Dec 17;13:1194. doi: 10.1186/1471-2458-13-1194. PMID 24341761
- [Background] Perret C, Poiraudeau S, Fermanian J, Colau MM, Benhamou MA, Revel M. Validity, reliability, and responsiveness of the fingertip-to-floor test. Arch Phys Med Rehabil. 2001 Nov;82(11):1566-70. doi: 10.1053/apmr.2001.26064. PMID 11689977
- [Background] Helou K, El Helou N, Mahfouz M, Mahfouz Y, Salameh P, Harmouche-Karaki M. Validity and reliability of an adapted arabic version of the long international physical activity questionnaire. BMC Public Health. 2017 Jul 24;18(1):49. doi: 10.1186/s12889-017-4599-7. PMID 28738790
- [Background] Kim Y, Park I, Kang M. Convergent validity of the international physical activity questionnaire (IPAQ): meta-analysis. Public Health Nutr. 2013 Mar;16(3):440-52. doi: 10.1017/S1368980012002996. Epub 2012 Jul 2. PMID 22874087
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Algarni AS, Ghorbel S, Jones JG, Guermazi M. Validation of an Arabic version of the Oswestry index in Saudi Arabia. Ann Phys Rehabil Med. 2014 Dec;57(9-10):653-63. doi: 10.1016/j.rehab.2014.06.006. Epub 2014 Aug 4. PMID 25262247
- [Background] Amundsen PA, Evans DW, Rajendran D, Bright P, Bjorkli T, Eldridge S, Buchbinder R, Underwood M, Froud R. Inclusion and exclusion criteria used in non-specific low back pain trials: a review of randomised controlled trials published between 2006 and 2012. BMC Musculoskelet Disord. 2018 Apr 12;19(1):113. doi: 10.1186/s12891-018-2034-6. PMID 29650015
- [Background] Naguib PR, Elsayaad MM, Mohamed HH, Lasheen YR. Efficacy of side lying traction versus supine lying traction in treatment of lumbar disc herniation: A randomized controlled trial
- [Background] Kumari A, Quddus N, Meena PR, Alghadir AH, Khan M. Effects of One-Fifth, One-Third, and One-Half of the Bodyweight Lumbar Traction on the Straight Leg Raise Test and Pain in Prolapsed Intervertebral Disc Patients: A Randomized Controlled Trial. Biomed Res Int. 2021 Sep 16;2021:2561502. doi: 10.1155/2021/2561502. eCollection 2021. PMID 34568490
- [Background] Kılıç Ç, Öz B, Ölmez N, Günay Uçurum S, Memiş A. Clinical and Functional Effects of Traction for Lumbar Disk Hernia Patients. Acta Med Nicomedia. February 2021;4(1):4-10.
- [Background] Khan RR, Riaz S, Rashid S, Sulman M. Effectiveness of mechanical traction in supine versus prone lying position for lumbosacral radiculopathy. Pak J Med Sci. 2021 Sep-Oct;37(5):1451-1455. doi: 10.12669/pjms.37.5.4200. PMID 34475929
- [Background] Thackeray A, Fritz JM, Childs JD, Brennan GP. The Effectiveness of Mechanical Traction Among Subgroups of Patients With Low Back Pain and Leg Pain: A Randomized Trial. J Orthop Sports Phys Ther. 2016 Mar;46(3):144-54. doi: 10.2519/jospt.2016.6238. Epub 2016 Jan 26. PMID 26813755
- [Background] Vanti C, Panizzolo A, Turone L, Guccione AA, Violante FS, Pillastrini P, Bertozzi L. Effectiveness of Mechanical Traction for Lumbar Radiculopathy: A Systematic Review and Meta-Analysis. Phys Ther. 2021 Mar 3;101(3):pzaa231. doi: 10.1093/ptj/pzaa231. PMID 33382419
- [Background] Wang W, Long F, Wu X, Li S, Lin J. Clinical Efficacy of Mechanical Traction as Physical Therapy for Lumbar Disc Herniation: A Meta-Analysis. Comput Math Methods Med. 2022 Jun 21;2022:5670303. doi: 10.1155/2022/5670303. eCollection 2022. PMID 35774300
- [Background] Vanti C, Saccardo K, Panizzolo A, Turone L, Guccione AA, Pillastrini P. The effects of the addition of mechanical traction to physical therapy on low back pain? A systematic review with meta-analysis. Acta Orthop Traumatol Turc. 2023 Jan;57(1):3-16. doi: 10.5152/j.aott.2023.21323. PMID 36939359
- [Background] Bilgilisoy Filiz M, Kilic Z, Uckun A, Cakir T, Koldas Dogan S, Toraman NF. Mechanical Traction for Lumbar Radicular Pain: Supine or Prone? A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Jun;97(6):433-439. doi: 10.1097/PHM.0000000000000892. PMID 29309314
- [Background] Cheng YH, Hsu CY, Lin YN. The effect of mechanical traction on low back pain in patients with herniated intervertebral disks: a systemic review and meta-analysis. Clin Rehabil. 2020 Jan;34(1):13-22. doi: 10.1177/0269215519872528. Epub 2019 Aug 28. PMID 31456418
- [Background] Gati T, Czimer E, Cserhati G, Feher J, Olah M, Kulisch A, Mando Z, Bender T. A multicentre randomized controlled follow-up study of the effects of the underwater traction therapy in chronic low back pain. Int J Biometeorol. 2020 Aug;64(8):1393-1400. doi: 10.1007/s00484-020-01919-8. Epub 2020 May 2. PMID 32361959
- [Background] Alrwaily M, Almutiri M, Schneider M. Assessment of variability in traction interventions for patients with low back pain: a systematic review. Chiropr Man Therap. 2018 Sep 17;26:35. doi: 10.1186/s12998-018-0205-z. eCollection 2018. PMID 30237870
- [Background] Wegner I, Widyahening IS, van Tulder MW, Blomberg SE, de Vet HC, Bronfort G, Bouter LM, van der Heijden GJ. Traction for low-back pain with or without sciatica. Cochrane Database Syst Rev. 2013 Aug 19;2013(8):CD003010. doi: 10.1002/14651858.CD003010.pub5. PMID 23959683
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Miftari S, Shukova Stojanovska D, Ismajli B, Rrecaj-Malaj S. The Effect of Combined Treatment with Passive Therapy, Physical Exercises, Lumbar Traction, and Walking Program on Chronic Low Back Pain. Sport Mont. 2023 Jun 1;21(2):97-101.
- [Background] Ibsen C, Maribo T, Nielsen CV, Horder M, Schiottz-Christensen B. ICF-Based Assessment of Functioning in Daily Clinical Practice. A Promising Direction Toward Patient-Centred Care in Patients With Low Back Pain. Front Rehabil Sci. 2021 Oct 26;2:732594. doi: 10.3389/fresc.2021.732594. eCollection 2021. PMID 36188866
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Jones M, Stratton G, Reilly T, Unnithan V. The efficacy of exercise as an intervention to treat recurrent nonspecific low back pain in adolescents. Pediatr Exerc Sci. 2007 Aug;19(3):349-59. doi: 10.1123/pes.19.3.349. PMID 18019593
- [Background] Alhakami AM, Davis S, Qasheesh M, Shaphe A, Chahal A. Effects of McKenzie and stabilization exercises in reducing pain intensity and functional disability in individuals with nonspecific chronic low back pain: a systematic review. J Phys Ther Sci. 2019 Jul;31(7):590-597. doi: 10.1589/jpts.31.590. Epub 2019 Jul 9. PMID 31417227
- [Background] Vanti C, Turone L, Panizzolo A, Guccione AA, Bertozzi L, Pillastrini P. Vertical traction for lumbar radiculopathy: a systematic review. Arch Physiother. 2021 Mar 15;11(1):7. doi: 10.1186/s40945-021-00102-5. PMID 33715638
- [Background] Bardin LD, King P, Maher CG. Diagnostic triage for low back pain: a practical approach for primary care. Med J Aust. 2017 Apr 3;206(6):268-273. doi: 10.5694/mja16.00828. PMID 28359011
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708
- [Background] Aldera MA, Alexander CM, McGregor AH. Prevalence and Incidence of Low Back Pain in the Kingdom of Saudi Arabia: A Systematic Review. J Epidemiol Glob Health. 2020 Dec;10(4):269-275. doi: 10.2991/jegh.k.200417.001. Epub 2020 Apr 24. PMID 32959606
- [Background] Frizziero A, Pellizzon G, Vittadini F, Bigliardi D, Costantino C. Efficacy of Core Stability in Non-Specific Chronic Low Back Pain. J Funct Morphol Kinesiol. 2021 Apr 22;6(2):37. doi: 10.3390/jfmk6020037. PMID 33922389
- [Background] Hashimoto Y, Matsudaira K, Sawada SS, Gando Y, Kawakami R, Sloan RA, Kinugawa C, Okamoto T, Tsukamoto K, Miyachi M, Naito H. Association between objectively measured physical activity and body mass index with low back pain: a large-scale cross-sectional study of Japanese men. BMC Public Health. 2018 Mar 9;18(1):341. doi: 10.1186/s12889-018-5253-8. PMID 29523128
- [Background] de Lira MR, de Mello Meziat-Filho NA, Silva GZM, Chaves TC. Efficacy of the cognitive functional therapy (CFT) in patients with chronic nonspecific low back pain: a study protocol for a randomized sham-controlled trial. Trials. 2022 Jul 4;23(1):544. doi: 10.1186/s13063-022-06466-8. PMID 35788240
- [Background] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979